CLINICAL TRIAL: NCT04738955
Title: Prospective, Observational and Cohort Clinical Research on Clinical Efficacy and Safety of Different Doses of Micafungin Sodium for Injection in Prevention and Treatment of Fungal Infection in Patients With Hematological Tumors
Brief Title: Efficacy and Safety of Micafungin for Injection in Prevention and Treatment of Fungal Infection in Hematological Tumors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Director of Department of Hematology, Shandong Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShandongPH12
Record Dates: First submitted 2021-01-16; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Hematological Tumors Patients With High Risk Factors of Invasive Fungal Disease
Keywords: hematological tumors; Invasive Fungal Disease
MeSH Terms: conditions — Hematologic Neoplasms; Invasive Fungal Infections | interventions — Micafungin

STUDY DESIGN:
Intervention Model Description: The patients will be randomized either low dose group or high dose group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High dose group (Experimental): micafungin sodium ≥ 200, ≤ 300 mg/time, once a day, intravenous drip
  Interventions: Drug: Micafungin Sodium

INTERVENTIONS:
Drug: Micafungin Sodium — micafungin sodium ≥ 100, <200mg/time, once a day, intravenous drip. Low dose group

SUMMARY:
This is a multi-center, prospective, open, observational and optimal clinical research to evaluate the clinical effectiveness and safety of different doses of micafungin sodium for injection in patients with hematological tumors.

DETAILED DESCRIPTION:
This is a multi-center, prospective, open, observational and optimal clinical research to evaluate the clinical effectiveness and safety of different doses of micafungin sodium for injection in patients with hematological tumors. Researchers screened suitable subjects according to the admission criteria, and after signing the informed consent form, micafungin sodium for injection was used for preventive or empirical treatment. During the treatment period, subjects who need to change the treatment plan due to uncontrollable infection or other reasons will withdraw from this research and the researchers will decide the follow-up treatment plan.All subjects were monitored for efficacy and safety according to the visit plan during the research.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, male or female
2. Patients with hematological tumors
3. Neutropenia: The absolute neutrophils count (ANC) in peripheral blood was 0.5×109/L or was expected to be ANC<0.5×109/L 48 hours later.
4. Fever: single measurement of oral temperature ≥ 38.3℃ (axillary temperature ≥ 38.0℃) or oral temperature ≥ 38.0℃ (axillary temperature ≥ 37.7℃) lasts for more than 1h
5. Patients with high risk factors of IFD (Invasive Fungal Disease), such as patients treated with allo-HSCT, patients with acute leukemia (including MDS) undergoing primary induction or rescue chemotherapy, patients with expected granulocytosis lasting more than 10 days, patients with severe granulocytosis or patients with severe aplastic anemia receiving antithymic globulin (ATG) therapy or HSCT therapy, etc.

Exclusion Criteria:

1. The patient is being treated with an antifungal drug
2. People who are known or suspected to be allergic to echinocandins
3. The infection is suspected to be caused by parasites, viruses or Mycobacterium tuberculosis.
4. Existing drug sensitivity results suggest that patients resistant to micafungin
5. Severe chronic liver disease with Child-Pugh grade C
6. Fever caused by tumor
7. Micafungin in the Treatment of Fungal Infections Caused by Cryptococcus, Zygomycetes and Trichospora that Are Ineffective
8. Removal of the central venous catheter can effectively relieve fever, and it is difficult to determine whether micafungin is effective or not.
9. Patients who were not considered suitable for the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
clinical efficacy | 14 days
  Breakthrough incidence of Invasive Fungal Infection (IFI), during prophylaxis use of micafungin

SECONDARY OUTCOMES:
Safety assessed by lab-test and adverse events | 30 days
  Incidence of adverse reactions in different dose groups of micafungin
Survival rate | 30 days
  IFD-related mortality

CONTACTS AND LOCATIONS:
Overall Officials: xin wang, MD, PHD, Study Chair — Shandong Provincial Hospital
Locations (1):
- Department of Hematology, Provincial Hospital Affiliated to Shandong University, Jinan, Shandong, China